CLINICAL TRIAL: NCT01114646
Title: Functional Status, Morbidity and Mortality in Cemented Versus Uncemented Hemiarthroplasty for Subcapital Hip Fractures: A Prospective Randomized Trial
Brief Title: Functional Status, Morbidity and Mortality in Cemented Versus Press-Fit Hemiarthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hartford Hospital (Other)
Collaborators: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 03001334HU; 124013 (Other: Hartford Hospital IRB)
Record Dates: First submitted 2010-04-29; First posted 2010-05-03 (Estimated); Results first posted 2018-08-07 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2013-03

CONDITIONS: Femoral Neck Fracture
Keywords: Hemiarthroplasty; Cemented; Press Fit; Mortality; Morbidity; Functional Status; Displaced femoral neck fracture
MeSH Terms: conditions — Femoral Neck Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cemented Hip Hemiarthroplasty (Other): This arm received a hemiarthroplasty with a cemented femoral prosthesis (VerSys LD/Fx, Zimmer, Warsaw, IN).
  Interventions: Device: Cemented Hip Hemiarthroplasty
- Press-Fit Hip Hemiarthroplasty (Experimental): This arm received a press-fit hemiarthroplasty (VerSys Beaded FullCoat, Zimmer, Warsaw, IN),
  Interventions: Device: VerSys Beaded FullCoat, Zimmer

INTERVENTIONS:
Device: Cemented Hip Hemiarthroplasty — The cemented femoral prosthesis is a VerSys LD/Fx, Zimmer, Warsaw, IN.
  Arms: Cemented Hip Hemiarthroplasty
Device: VerSys Beaded FullCoat, Zimmer — The press-fit component is a VerSys Beaded FullCoat, Zimmer, Warsaw, IN,
  Arms: Press-Fit Hip Hemiarthroplasty

SUMMARY:
Hemiarthroplasty (half of a hip replacement) is the most common treatment for displaced fractures of the femoral neck in the elderly and is associated with a better functional outcome and fewer reoperations than internal fixation. Currently, the operative management of displaced femoral neck fractures favors the use of cemented implants. This technique is believed to be more stable in the immediate post-operative period, but there is limited evidence of a decreased morbidity and mortality with cemented versus press-fit stems (uncemented). In 2006, a meta-analysis concluded that the evidence was too limited to recommend a cemented or press-fit hemiarthroplasty.

In this investigation, the morbidity, mortality and functional outcome associated with cemented and press-fit hemiarthroplasty will be compared prospectively. We propose that the use of press-fit hemiarthroplasty in the treatment of displaced subcapital fractures of the femoral neck would be associated with a decreased risk of adverse peri-operative outcomes, and that the functional results of cemented and press-fit hemiarthroplasty will be equivalent at one year.

ELIGIBILITY:
Inclusion Criteria:

* older than 55 years
* non-pathologic, displaced subcapital femoral neck fracture
* designated for surgical reconstruction with a hemiarthroplasty by the attending surgeon
* able to ambulate ten feet prior to presentation

Exclusion Criteria:

* unable to walk ten feet prior to hip fracture
* multiple extremity trauma
* pathologic fracture of the hip (including malignancy)
* clinically recognized acute myocardial infarction within thirty days prior to enrollment
* previously participated in the trial
* symptoms associated with anemia
* pre-existing metabolic bone disease

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2005-03; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph P. DeAngelis, MD, Study Director — Hartford Hospital; Courtland G. Lewis, MD, Principal Investigator — Hartford Hospital
Locations (1):
- Hartford Hospital, Hartford, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cemented Hip Hemiarthroplasty | Press-Fit Hip Hemiarthroplasty
Started | 66 | 64
Completed | 63 | 62
Not Completed | 3 | 2
Not completed — Withdrawal by Subject | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cemented Hip Hemiarthroplasty | Press-Fit Hip Hemiarthroplasty | Total
Number analyzed (Participants) | 66 | 64 | 130
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 66 | 64 | 130
Age, Continuous [Mean (Standard Deviation); unit: years] | 81.8 (9.0) | 82.8 (7.6) | 82.3 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 48 | 100
  Male | 14 | 16 | 30
Region of Enrollment [Number; unit: participants]
  United States | 66 | 64 | 130

OUTCOME MEASURES:

1. Primary Outcome: Mortality
Description: Assessment of post-operative mortality at one-year.
Time Frame: 1 year
Measure: Number; unit: pecent
Arm/Group | Cemented Hip Hemiarthroplasty | Press-Fit Hip Hemiarthroplasty
Number analyzed (Participants) | 66 | 64
pecent | 23.1 | 20.1

2. Primary Outcome: Post-Operative Unstable Angina
Description: Unstable angina was defined as the new onset of prolonged chest pain (greater than or equal to 30 minutes) or two episodes of chest pain thought to be of cardiac origin or an electrocardiogram showing new T-wave inversion, ST depression or elevation with enzymes non-diagnostic of myocardial ischemia.
Time Frame: 1 week post-operation
Reporting Status: Not Posted

3. Primary Outcome: Post-Operative Myocardial Infarction
Description: Myocardial infarction required a positive troponin or electrocardiogram consistent with definite infarction.
Time Frame: 1 week post-operation
Reporting Status: Not Posted

4. Secondary Outcome: Instrumental Activities of Daily Living (IADL) and Physical Activities of Daily Living (PADL) Scale
Description: A modified version of the Older Americans Resources and Services Instrument (OARS) which asks about performance of tasks of daily living during the preceding two weeks.14 These activities include: getting to places, walking distances, shopping for groceries or clothes, preparing meals and doing housecleaning.
Time Frame: 1 year
Reporting Status: Not Posted

5. Secondary Outcome: Energy/Fatigue Scale
Description: An inquire about fatigue, level of energy and self-efficiency.
Time Frame: 1 year
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Post-randomization unstable angina, MI during the index hospitalization or death for any reason within 30 days.
Description: other events such pneumonia, wound infection, thromboembolic event, cerebrovascular accident major hemorrhage will be assessed by concurrent medical record review. Hospital outcome will be assessed by surgical and medical team. Functional outcome will be completed over the telephone (self-reported)
Arm/Group | Cemented Hip Hemiarthroplasty | Press-Fit Hip Hemiarthroplasty
Serious Adverse Events (participants affected / at risk) | 1/66 | 1/64
Other Adverse Events (participants affected / at risk) | 11/66 | 8/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cemented Hip Hemiarthroplasty (N=66) | Press-Fit Hip Hemiarthroplasty (N=64)
Death (Cardiac disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cemented Hip Hemiarthroplasty (N=66) | Press-Fit Hip Hemiarthroplasty (N=64)
ICU stay (General disorders) | 4 | 5
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Myocardial Infarction (Cardiac disorders) | 2 | 1
Wound Infection (Infections and infestations) | 1 | 1
Re-operation (Surgical and medical procedures) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No